CLINICAL TRIAL: NCT01089231
Title: Effects of Omega-3 Fatty Acids From Fish Oil on the Gene Expression in Healthy Humans and Humans With Hypertriglyceridemia
Brief Title: Effects of Omega-3 Fatty Acids on the Human Gene Expression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gottfried Wilhelm Leibniz Universität Hannover (Other)
Responsible Party: Principal Investigator, M. Sc. Simone Schmidt, Master of Science, Gottfried Wilhelm Leibniz Universität Hannover
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWLUH-001; GWLUH2010 (Other: 01)
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Hyperlipidemia; Healthy
Keywords: Hyperlipidemia; coronary heart disease; gene expression; fish oil; DHA, EPA
MeSH Terms: conditions — Hyperlipidemias; Coronary Disease | interventions — Fish Oils; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo - healthy subjects (Placebo Comparator): Dietary Supplement: corn oil capsules (6 per day) about 3 months
  Interventions: Dietary Supplement: Placebo (corn oil)
- Placebo - hyperlipedemic subjects (Placebo Comparator): Dietary Supplement: corn oil capsules (6 per day) about 3 months
  Interventions: Dietary Supplement: Placebo (corn oil)
- Fish oil - hyperlipidemic subjects (Experimental): Dietary Supplement: fish oil capsules (6 per day) 3024 mg n-3 fatty acids daily (1512 mg EPA and 1008 mg DHA) about 3 months
  Interventions: Dietary Supplement: Fish oil
- Fish oil - healthy subjects (Experimental): Dietary Supplement: fish oil capsules (6 per day) 3024 mg n-3 fatty acids daily (1512 mg EPA and 1008 mg DHA) about 3 months.
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil — Dietary Supplement: fish oil capsules (6 per day) 3024 mg n-3 fatty acids daily (1512 mg EPA and 1008 mg DHA) about 3 months
  Arms: Fish oil - healthy subjects; Fish oil - hyperlipidemic subjects
Dietary Supplement: Placebo (corn oil) — corn oil (6 capsules per day)
  Arms: Placebo - healthy subjects; Placebo - hyperlipedemic subjects

SUMMARY:
The aim of this study is to investigate the effects of short- and long-term intervention with EPA and DHA-rich fish oil on gene expression profiles in healthy and hyperlipidemic males.

DETAILED DESCRIPTION:
Cardiovascular and coronary heart diseases continue to be the leading causes of morbidity and mortality among adults in Europe and North America. Since the number of elderly people and therefore the number of chronic-inflammatory diseases rise, preventive therapies become more important. Within preventive strategies, nutrition plays a central role.

Cross-sectional studies suggested that omega-3 fatty acids, especially the very long-chain fatty acids Eicosapentaenoic acid (EPA, C20:5ω3) and Docosahexaenoic acid (DHA, C22:6ω3), are protective against cardiovascular and coronary heart diseases. Their cardio protective potential is based on their positive effects on blood lipids, vascular tonus and blood clotting. A number of controlled clinical trials have shown that EPA and DHA supplementation lower fasting and postprandial plasma concentrations of triglyceride-rich lipoproteins and their remnants. Biochemical research revealed numerous metabolic effects of EPA and DHA, ranging from their effects on membrane fluidity to the modification of the eicosanoid profile.

However, only a few human clinical trials examined the regulative effects of DHA and EPA supplementation on gene expression. Furthermore, to our knowledge no published research data is available dealing with the effect of these fatty acids on gene expression in subjects with hypertriglyceridemia in comparison to healthy subjects. Such findings are of great concern due to hints that especially people with hypertriglyceridemia benefit from the triglyceride lowering effect of EPA and DHA supplementation. Presently it is not well-established if the gene regulative potential of EPA and DHA in these persons differs from healthy persons. These findings could help to understand the differences in the metabolic effects of EPA and DHA in healthy vs. hypertriglyceridemic persons, which have a greater risk for cardiovascular and coronary diseases. Finally, these data could contribute to a knowledge basis for targeted strategies in preventive therapies with the very long-chain omega-3 fatty acids EPA and DHA.

ELIGIBILITY:
Inclusion Criteria:

* males, 20-50 years
* non-smokers
* ethnicity: Caucasians
* no medical treatment
* healthy subjects:

  * no documented disease
  * normal blood lipids (triglyceride < 150 mg/dl; total cholesterol < 200 mg/dl)
* humans with increased blood lipids (hyperlipidemia)

  * documented hypertriglyceridemia or
  * triglyceride ≥ 150 mg/dl (≥ 1,7 mmol/l) and
  * total cholesterol > 200 mg/dl (5,2 mmol/l)
* written confirmation of the subjects after detailed oral and written explanation about the study contents, - requirements and risks
* ability and willingness of the participants to attend the investigator's orders (compliance of the study conditions, consumption of the study medicaments according to the dosage commendation)

Exclusion Criteria:

* Body-Mass-Index (BMI) ≥ 35
* smokers
* medical treatment (especially corticosteroids, anti-inflammatory drugs, blood lipids lowering drugs (e.g. statins, fibrates, bile acid exchanger resin, phytosterols)
* taking any supplements with omega-3 fatty acids, phytosterols, polyglucosamines (Chitosan) or other lipid binding ingredients
* daily consumption of omega-3 fatty acids rich fish (salmon, mackerel, herring)
* heavy chronic diseases (tumors, diabetes typ 1, etc.), documented heart disease, documented blood clotting disorders, renal failure, liver diseases
* documented blood clotting disorders and consumption of coagulation-inhibiting drugs (for example Marcumar, ASS)
* allergy or intolerance to fish/fish oil or any of the study ingredients of the test products
* chronic gastro-intestinal diseases (Colitis ulcerosa, Morbus Crohn, pancreatic insufficiency)
* donation of blood in the last 6 weeks
* routine consumption of laxative
* common exclusion criteria like

  * alcohol-, drug- and/or medicament dependence
  * subjects who are not in agreement with the study conditions
  * refusal or rather reset of the consent from the subject
  * active participation in other investigational drug or device trial within the last 30 days

Ages: 20 Years to 51 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hahn, Prof., Study Director — Gottfried Wilhelm Leibniz University of Hanover
Locations (1):
- Gottfried Wilhelm Leibniz University of Hanover, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Schmidt S, Willers J, Stahl F, Mutz KO, Scheper T, Hahn A, Schuchardt JP. Regulation of lipid metabolism-related gene expression in whole blood cells of normo- and dyslipidemic men after fish oil supplementation. Lipids Health Dis. 2012 Dec 14;11:172. doi: 10.1186/1476-511X-11-172. PMID 23241455
- [Derived] Schmidt S, Stahl F, Mutz KO, Scheper T, Hahn A, Schuchardt JP. Different gene expression profiles in normo- and dyslipidemic men after fish oil supplementation: results from a randomized controlled trial. Lipids Health Dis. 2012 Aug 29;11:105. doi: 10.1186/1476-511X-11-105. PMID 22929118
- [Derived] Schmidt S, Stahl F, Mutz KO, Scheper T, Hahn A, Schuchardt JP. Transcriptome-based identification of antioxidative gene expression after fish oil supplementation in normo- and dyslipidemic men. Nutr Metab (Lond). 2012 May 23;9(1):45. doi: 10.1186/1743-7075-9-45. PMID 22621246
- See also: web page of the institute — http://www.nutrition.uni-hannover.de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of subjects was performed by several advertisements and study placards in hanover from january until february 2010. By a telephonic preselection 106 subjects were selected according to inclusion criteria.
Pre-assignment Details: Serum lipid levels of the preselected subjects were determined and 20 normolipidemic and 20 dyslipidemic men were enrolled in the study population.
Groups:
- Placebo - Healthy Subjects: Dietary Supplement: corn oil capsules (6 per day) about 3 months n=6
- Placebo - Hyperlipedemic Subjects: Dietary Supplement: corn oil capsules (6 per day) about 3 months n=8
- Fish Oil - Hyperlipidemic Subjects: Dietary Supplement: fish oil capsules (6 per day) 3024 mg n-3 fatty acids daily (1512 mg EPA and 1008 mg DHA) about 3 months n=8
- Fish Oil - Healthy Subjects: Dietary Supplement: fish oil capsules (6 per day) 3024 mg n-3 fatty acids daily (1512 mg EPA and 1008 mg DHA) about 3 months. n=9
Period: Overall Study
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects
Started | 10 | 10 | 10 | 10
Completed | 6 (4 subjects excluded (2 alcohol use / TG level changes; 1 use of not allowed drugs; 1 low RNA yield)) | 8 (2 subjects excluded (1 highly elevated TG and TC data; 1 elevated inflammation (CRP level))) | 8 (2 subject excluded (1 use of not allowed drugs; 1 low RNA yield)) | 9 (1 subject excluded (low RNA yield))
Not Completed | 4 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.4 (8.30) | 41.8 (8.94) | 40.2 (8.64) | 37.5 (8.11) | 38.82 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 10 | 40
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Gene Expression Changes
Description: Gene expression changes were measured by using whole genome microarrays. The expression values of all genes were compared between baseline and 4 hours, 7 days and twelve weeks after supplementation with FO or CO and differentially expressed genes were detected by standard two-state pooled-variance t-test (p<0,05). The number of differentially expressed genes (regulated genes)compared to the baseline values were determined for every study group in total as well as for every time point (4 hours, 7 days, 12 weeks)in total and specifically.
Time Frame: Gene expression changes (number of regulated genes)
Measure: Number; unit: number of regulated genes
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects
Number analyzed (Participants) | 6 | 8 | 8 | 9
number of regulated genes
  total (4 hours+7 days+12weeks,without doubles) | 841 | 1041 | 1639 | 628
  4 hours (total) | 320 | 436 | 508 | 264
  7 days (total) | 418 | 629 | 1105 | 230
  12 weeks (total) | 500 | 493 | 1027 | 338
  4 hours (specific) | 94 | 85 | 246 | 140
  7 days (specific) | 135 | 242 | 326 | 78
  12 weeks (specific) | 312 | 287 | 203 | 214

2. Secondary Outcome: Fatty Acid Composition of Erythrocyte Membranes (Omega-3 Index)
Description: Fasting venous blood samples were collected and RBC membrane FA composition including the omega-3 index, given as EPA + DHA, was analyzed at baseline and after 12 weeks according to the omega-3 index methodology (Harris & von Schacky, 2004). Results are presented as a percentage of the total identified FAs after response factor correction. The coefficient of variation for EPA + DHA was 5%. Quality was assured according to DIN ISO 15189.
Time Frame: baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total fatty acids
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects
Number analyzed (Participants) | 6 | 8 | 8 | 9
percentage of total fatty acids
  omega-3 index baseline | 5.08 (1.41) | 5.27 (1.69) | 4.90 (1.80) | 5.24 (0.70)
  omega-3 index after 12 weeks | 4.78 (1.16) | 5.50 (1.57) | 9.84 (1.26) | 10.7 (1.06)

3. Secondary Outcome: Blood Lipids
Description: Fasting venous blood samples were collected and blood lipid levels were determined by an external contract laboratory (LADR, Hannover; Germany) at baseline (t0), after one week (t1) and after 12 weeks (t12) of supplementation.
Time Frame: baseline and after 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects
Number analyzed (Participants) | 6 | 8 | 8 | 9
mg/dl
  total cholesterol (TC) baseline | 194.0 (22.2) | 261.0 (48.1) | 262.2 (61.9) | 184.1 (13.3)
  total cholesterol (TC) after 12 weeks | 188.9 (21.5) | 257.5 (60.3) | 264.4 (49.2) | 198.6 (26.1)
  low-density lipoprotein (LDL) baseline | 118.1 (25.1) | 178.1 (45.4) | 146.1 (5.31) | 108.7 (12.8)
  low-density lipoprotein (LDL) after 12 weeks | 118.6 (28.2) | 172.6 (54.4) | 167.4 (23.6) | 117.2 (22.1)
  high-density lipoprotein (HDL) baseline | 52.7 (12.7) | 47.9 (10.0) | 45.2 (6.5) | 59.0 (10.4)
  high-density lipoprotein (HDL) after 12 weeks | 52.6 (11.6) | 47.4 (8.21) | 50.8 (9.43) | 65.2 (14.4)
  triacylglycerol (TG) baseline | 115.6 (53.8) | 175.0 (56.2) | 322.4 (259.0) | 82.4 (35.3)
  triacylglycerol (TG) after 12 weeks | 87.4 (14.8) | 186.9 (49.6) | 230.8 (147.0) | 66.2 (16.7)

ADVERSE EVENTS:
Arm/Group | Placebo - Healthy Subjects | Placebo - Hyperlipedemic Subjects | Fish Oil - Hyperlipidemic Subjects | Fish Oil - Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
* A higher number of participants would be better to compensate drop outs
* two pre-screening procedures of lipid levels are generally desirable
* CO is not an optimal placebo control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No